CLINICAL TRIAL: NCT02723227
Title: The Impact of Family Financial Support on Parental Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adam Schickedanz, Clinical Instructor in Pediatrics and Clinical Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLASchickedanzFCS
Record Dates: First submitted 2016-03-25; First posted 2016-03-30 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Stress
Keywords: Parenting Stress; Stress; Social Determinants; Socioeconomic status; Financial Coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial Coaching & Social Service Referral (Experimental): Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Interventions: Behavioral: Financial Coaching; Behavioral: Referral to Social Services
- Social Services Referral (Active Comparator): Enrollment provides for access to referrals to social services.
  Interventions: Behavioral: Referral to Social Services

INTERVENTIONS:
Behavioral: Financial Coaching — Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Arms: Financial Coaching & Social Service Referral
Behavioral: Referral to Social Services

SUMMARY:
The investigators have partnered with financial coaching organizations to establish what the investigators have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on family economic strain and parental stress.

DETAILED DESCRIPTION:
Financial coaching is a new tool in the field of community development, but it has already demonstrated significant financial impact in a number of studies, including one randomized trial conducted by the Urban Institute. Financial coaching improves participant financial literacy, budgeting, saving for financial emergencies, and debt level. The investigators' project will help clinicians and the field of community economic development understand health and well-being through a new economic lens and assess the health-related impacts of the emerging field of financial coaching. The investigators have partnered with financial coaching organizations to establish what they have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on parental strain and stress.

Community-based participants will be recruited from South Los Angeles and randomized to receive either monthly financial coaching plus access to referral for social services (intervention) or access to referral for social services alone (control). Inclusion criteria include having dependents under age 18, having some form of income, and having a tax identification number (social security number or Individual Tax Identification Number). Participants will be surveyed quarterly regarding their economic strain using the Family Economic Strain Scale and their individual stress using the Parenting Stress Index.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include caregivers and parents with one or more dependents, some form of income, and a tax identification number.

Exclusion Criteria:

* Inability to partake in the financial coaching or primary language other than English or Spanish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Family Economic Strain | Up to one year (if possible)
  Parents will be asked to assess the degree to which their economic circumstances impact their family functioning using the Family Economic Strain Scale
Parenting Stress | Up to one year (if possible)
  Parents will be asked to quantify their parenting stress using the Parenting Stress Index

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schickedanz, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- LIFT-LA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participant consent did not include data sharing and there is no appropriate repository to share data with